CLINICAL TRIAL: NCT04846400
Title: Pilot Study of Novel Nasopharyngeal Airway Device for Treating Upper Airway Obstruction in Pediatric Hypotonia
Brief Title: Pilot Study of a Self-Supporting Nasopharyngeal Airway in Hypotonia
Acronym: ssNPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Zopf, Assistant Professor of Otolaryngology-Head and Neck Surgery, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R61HL151952 (NIH); R61HL151952 (NIH)
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Results first posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Sleep Apnea, Obstructive; Hypotonia; Child, Only
Keywords: Obstructive sleep apnea; Hypotonia; Nasal airway; Tolerability
MeSH Terms: conditions — Sleep Apnea, Obstructive; Muscle Hypotonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- ssNPA (Experimental): self-supporting nasopharyngeal airway to be used nightly for approximately 8 weeks.
  Interventions: Device: ssNPA

INTERVENTIONS:
Device: ssNPA — The ssNPA is a self-supporting nasopharyngeal airway, a stent that is a non-surgical alternative to treat severe OSA

SUMMARY:
Children with hypotonic upper airway obstruction have a high prevalence of severe obstructive sleep apnea, which if not treated has significant clinical consequence. Available treatment approaches, such as surgery and positive airway pressure, show limited efficacy and adherence. The multidisciplinary team has developed and now proposes to further test a non-surgical, well-tolerated nasopharyngeal airway device that in initial patients has resolved even extremely severe obstructive sleep apnea, and improved patient and family quality of life.

DETAILED DESCRIPTION:
There is a critical need for safe and effective treatment options for persistent obstructive sleep apnea (OSA) in patients with Hypotonic Upper Airway Obstruction (HUAO). HUAO encompass conditions such as cerebral palsy, hypoxic encephalopathy, syndromic tone anomalies, and neuromuscular disorders, and typically share a similar pattern of multisite upper airway collapse. OSA is characterized by recurrent episodes of partial or complete upper airway obstruction during sleep with associated arousals and/ or oxygen desaturations. Of hypotonic patients with symptoms of sleep disordered breathing, one quarter have moderate OSA, and more than half have severe OSA. Thus, not only are patients more likely to have OSA, but it is likely to be much more severe. Currently available treatment options, ranging from palliative care to tracheostomy, often fail to fully meet the needs of these patients. The multidisciplinary team has developed a dramatically effective non-surgical nasopharyngeal airway stent that has demonstrated good tolerability in hypotonic patients. This initial phase will test an enhanced version of the device for acceptability and tolerability. Critically, insertion, adherence, and compliance protocols will be optimized for preparation of the full trial.

This record originally included the Secondary Outcome Measure "Device Design". This Secondary Outcome Measure was removed during the results reporting process upon advisement of ClinicalTrials.gov reviewers, as it was not a directly health-related outcome.

ELIGIBILITY:
Inclusion Criteria:

* Children with HUAO: This includes those who newly diagnosed with OSA. These children will undergo overnight polysomnography to determine the presence of OSA (AHI>10 or AHI>5 with nocturnal hypoxemia defined as SpO2 nadir <=75%).
* Obstructive sleep apnea on polysomnogram with AHI>=10
* Presence of at least one symptom of OSA (such as snoring 3 or more nights per week, daytime sleepiness, or hyperactive/inattentive behaviors)
* Post adeonotonsillectomy or those with contraindications to tonsillectomy.
* obstructive sleep apnea on polysomnogram with AHI>=10
* Tonsil size 2+ or smaller
* Parent/caregivers willing and able to provide informed consent and child willing and able to provide assent, where appropriate.

Exclusion Criteria:

* AHI ≤10 on polysomnogram without hypoxemia or AHI<5 with hypoxemia - any reason why ssNPA may not be suitable
* Any medical reason why ssNPA therapy may not be suitable
* Active COVID 19 infections
* ETCO2 or TCO2 values >60 mmHg for >10% of sleep time on PSG
* Psychiatric, medical, or social factors likely to invalidate assessments, make adherence with ssNPA highly unlikely or make local follow-up at 8 weeks unfeasible. Some psychiatric conditions may be provoked or exacerbated by OSA, and those most commonly implicated - Attention Deficit/Hyperactivity Disorder, Conduct Disorder, and Oppositional Defiant Disorder - will not be exclusions. However, more pervasive conditions such as severe autism will be excluded
* Presence of supraglottic airway collapse or more distal airway stenosis or collapse (for example glottic, subglottic stenosis, or concern for distal airway stenosis or malacia)
* Moderate/severe tracheobroncomalacia
* Need for anticoagulative therapy
* Bleeding disorder
* Restrictive thoracic disorders

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Zopf, MD, Principal Investigator — University of Michigan
Locations (1):
- C.S. Mott Children's Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
For this initial pilot of 5 participants there are no plans to share data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ssNPA
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ssNPA
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Ability to Tolerate Measured by Percent of Participants With Protocol Goal
Description: Protocol objective was to achieve a score of >=7 in at least 60% of participants. Score of >=7 on Likert scale 0-10 (higher score is better).
Time Frame: 8 weeks
Measure: Number; unit: percent of participants
Arm/Group | ssNPA
Number analyzed (Participants) | 2
percent of participants | 50

2. Primary Outcome: Comfort as Measured by Percent of Participants With Protocol Objective Score
Description: Protocol objective was to achieve a score of >=6 in at least 60% of participants. Score of >=6 on Likert scale 0-10 (higher score is better).
Time Frame: 8 weeks
Measure: Number; unit: percent of participants
Arm/Group | ssNPA
Number analyzed (Participants) | 2
percent of participants | 100

3. Primary Outcome: Ease of Use as Indicated by Percent of Participants Whose Parents Responded Favorably to Device Use, With Protocol Goal
Description: Score of >=5 on Likert scale 1-10 (higher score is better).
Time Frame: 8 weeks
Measure: Number; unit: percent of participants
Arm/Group | ssNPA
Number analyzed (Participants) | 2
percent of participants | 100

4. Secondary Outcome: Snoring
Description: Less frequent snoring, as measured by scores of 1 or 2 on a question that read: While using the device my child's snoring occurred:
  1 much less often; 2: less often; 3: unchanged; 4: more often; 5: much more
Time Frame: 8 weeks
Population: One participant was an inconsistent user of the device, therefore 8 week survey data is not available. Since Clinicaltrials.gov's purpose is not to show individual level results, the results for the consistent user are not shown here.
Arm/Group | ssNPA
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Daytime Sleepiness as Shown by Number of Participants Who Had a Reduction in Their Epworth Sleepiness Scale Score
Description: Reduction in Epworth Sleepiness Scale score (0-24; lower score is better);
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ssNPA
Number analyzed (Participants) | 2
Participants | 1

6. Secondary Outcome: Sleep Quality, as Measured by Number of Participants With Parent Identified Improved Sleep
Description: Number of participants whose parents' response on the sleep quality improvement question were >=7. Change in sleep quality was reported on a 1-10 scale, where 1 was greatest worsening of sleep and 10 was most improved sleep.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ssNPA
Number analyzed (Participants) | 2
Participants | 2

7. Secondary Outcome: Insertion Protocol Optimization as Measured by Percent of Participants Who Found Insertion Relatively Easy
Description: Percent of participants who reported a score of <= 5 on Likert scale of 1-10, where lower score indicates easier insertion.
Time Frame: 8 weeks
Measure: Number; unit: percent of participants
Arm/Group | ssNPA
Number analyzed (Participants) | 2
percent of participants | 100

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | ssNPA
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT04846400/Prot_SAP_001.pdf